CLINICAL TRIAL: NCT05719337
Title: Characteristics of the Multi-Modality Echocardiographic Techniques in Chinese Adults With Pathological Left Ventricular Hypertrophy - a Prospective, Multicenter, Clinical Study (MET-LVH Study)
Brief Title: Multi-Modality Echocardiographic Techniques in Pathological Left Ventricular Hypertrophy Adults
Acronym: MET-LVH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Hospital of China Medical University (Other)
Collaborators: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Chunyan Ma, Chief of Cardiovascular Ultrasound, First Hospital of China Medical University
Other Study IDs: MET-LVH-01
Record Dates: First submitted 2023-01-29; First posted 2023-02-08 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Left Ventricular Hypertrophy
Keywords: Pathological Left Ventricular Hypertrophy; Multi-modality Echocardiographic Parameters; Hypertensive Heart Disease; Hypertrophic Cardiomyopathy; Cardiac Amyloidosis; Fabry Disease
MeSH Terms: conditions — Hypertrophy, Left Ventricular; Cardiomyopathy, Hypertrophic; Amyloid Neuropathies, Familial; Fabry Disease | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Hypertensive heart disease group: Systolic blood pressure exceeded 140 mmHg and/or diastolic blood pressure exceeded 90 mmHg, or a history of systemic hypertension in the absence of other cardiac or systemic disease was described as hypertension.
  Interventions: Device: Echocardiography
- Hypertrophic cardiomyopathy group: Wall thickness≥15 mm in the absence of other causes of hypertrophy in a non-dilated left ventricle (LV) defines HCM. End diastolic wall thickness≥13 mm can be diagnostic if there is a family history of HCM or a known disease-causing genetic mutation.
  Interventions: Device: Echocardiography
- Cardiac amyloidosis group: Clinical diagnosis of cardiac amyloidosis confirmed by blood tests or tissue biopsy.
  Interventions: Device: Echocardiography
- Fabry disease group: Clinical diagnosis of Fabray disease confirmed by blood biomarkers or genetic testing.
  Interventions: Device: Echocardiography

INTERVENTIONS:
Device: Echocardiography — Two-dimensional, color Doppler, spectral Doppler, tissue Doppler and three-dimensional echocardiographic image recordings will be taken using a Philips Epiq 7C echocardiography device and X5-1 probe. Conventional parameters, additional parameters, and strain analyzes will be performed by TomTec AutoStrain Suite Software.

SUMMARY:
This multicenter clinical study aims to evaluate the multi-modality echocardiographic parameters in patients with different pathological left ventricular hypertrophy (LVH) and investigate the correlation between echocardiographic parameters and different etiologies, providing an important theoretical basis for early identification and risk assessment in LVH patients.

DETAILED DESCRIPTION:
Left ventricular hypertrophy (LVH) is an abnormal increase in the mass of the left ventricular myocardium, and its presence is associated with poor outcomes and ventricular arrhythmias. It is commonly seen in hypertension and aortic stenosis due to persistent pressure overload. In addition, it can also be found in genetic diseases and metabolic diseases, such as hypertrophic cardiomyopathy, cardiac amyloidosis and Fabry disease. Although patients with the latter type of LVH may often have normal loading conditions, there is significant heterogeneity in phenotypes and prognosis due to etiological variability. Hence for LVH patients, early identification of the underlying causes, effective intervention, follow up and surveillance may reduce mortality and improve survival. Echocardiography is the initial imaging modality for evaluation of cardiovascular diseases. And it plays an important role in the detection of LVH and potential causes in current clinical practice. Nevertheless, the feasibility of discriminatory for different diseases is limited by the fact that overlapping LVH in different conditions can often lead to diagnostic ambiguity. There is an urgent need to find echocardiographic parameters with high specificity to assist in the etiological diagnosis of patients with pathological LVH.

Patients with LVH commonly associate with left ventricular diastolic dysfunction, causing changes in the structure and function of the left atrium prior to abnormal left ventricular ejection fraction. Left atrium function at reservoir, conduit and booster phases can be noninvasively quantify by speckle tracking echocardiography. However, there is incomplete information on left atrium strain characteristics in patients with LV pathological hypertrophy. The myocardial longitudinal strain parameters derived from speckle tracking echocardiography is a sensitive noninvasive method of assessing left ventricular myocardial performance. The relative "apical sparing" can be easily visualized for patients with cardiac amyloidosis. The reduced longitudinal strain in the basal lateral wall could be found at the very early stages of Fabry disease. Hence the specific manifestations derived from longitudinal strain mapping can assist in the differentiate patients from various causes of LVH. And left ventricular volume and mass index assessed by three-dimension echocardiography are independently associated with adverse outcomes of LVH patients. Therefore, appropriate utilization of multi-modality echocardiography techniques is fundamental to accurate diagnosis as well as longitudinal care of pathological LVH patients. However, a great deal of studies were based on small samples and single center. There is lack of defined diagnostic results based on multi-modality echocardiography and comprehensive markers derived from large-scale study.

In this study, we expected to provide a set of parameters for different etiology by including patients with different pathological LVH based on multi-modality echocardiography, so as to assisting in early identification and risk assessment in LVH patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old;
* A wall thickness ≥ 12mm in one or more LV myocardial segments as measured by 2D echocardiography.
* Patients with definite diagnosis of hypertensive heart disease, hypertrophic cardiomyopathy, cardiac amyloidosis or Fabry disease.

Exclusion Criteria:

* Patients with severe valvular disease, congenital heart disease, aortic coarctation, multiple Takayasu arteritis, or other cardiovascular diseases that may cause ventricular hypertrophy;
* Hypertrophy of myocardium caused by high intensity exercise;
* Poor ultrasonic image quality, which cannot meet analysis requirement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with left ventricular hypertrophy (LVH) detected by echocardiography.
Sampling Method: Probability Sample
Enrollment: 660 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-08-05 (Estimated); Study Completion 2025-08-05 (Estimated)

PRIMARY OUTCOMES:
Conventional echocardiographic parameters in all pathological LVH patients | 1 day after admission
  To evaluate the conventional two-dimensional, color Doppler, spectral Doppler and tissue Doppler echocardiographic parameters in all pathological LVH patients.

SECONDARY OUTCOMES:
Strain parameters in all pathological LVH patients | 1 day after admission
  To evaluate the two-dimensional strain parameters of left ventricular and left atrium in all LVH patients.
Volume and mass parameters in all pathological LVH patients | 1 day after admission
  To evaluate the three-dimensional volume and mass parameters in all LVH patients.

CONTACTS AND LOCATIONS:
Overall Officials: Chunyan Ma, Ph.D, Principal Investigator — the First Hospital of China Medical Univeristy; Li Zhang, Ph.D, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (22):
- China (22):
  - the Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - the First Affiliated Hospital of Jiamusi University, Jiamusi, Heilongjiang
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - the Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Ansteel Group General Hospita, Anshan, Liaoning
  - Benxi Central Hospital, Benxi, Liaoning
  - Chaoyang Central Hospital, Chaoyang, Liaoning
  - Dalian Municipal Central Hospital, Dalian, Liaoning
  - the Second Hospital of Dalian Medical University, Dalian, Liaoning
  - Dandong Central Hospital, Dandong, Liaoning
  - Fushun Central Hospital, Fushun, Liaoning
  - the First Affiliated Hospital of Jinzhou Medical University, Jinzhou, Liaoning
  - Affiliated Central Hospital of Shenyang Medical College, Shenyang, Liaoning
  - Dadong Branch of First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - the First Affiliated Hospital of Liaoning University of Traditional Chinese Medicine, Shenyang, Liaoning
  - the First Hospital of China Medical Univeristy, Shenyang, Liaoning
  - the Second Affiliated Hospital of Shenyang Medical College, Shenyang, Liaoning
  - Liao Jian Group Tie Mei General Hospital, Tieling, Liaoning
  - Tieling Central Hospital, Tieling, Liaoning
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Undecided